CLINICAL TRIAL: NCT05828134
Title: Enhancing Muscle Health and Metabolism in Pre-frail Middle-aged and Older Adults: A Randomized Controlled Trial Investigating the Benefits of Protein-enriched Supplementation and Weekly Exercise
Brief Title: Enhancing Muscle Health and Metabolism in Pre-frail Middle-aged and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Laurel Enterprises Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YM109172F
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-04

CONDITIONS: Muscle Loss; Muscle Weakness
Keywords: Laurel Corporation; Protein-Enriched Soup
MeSH Terms: conditions — Muscular Atrophy; Muscle Weakness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care group (No Intervention): The control group only performed routine data collection and gave them dietary suggestion.
- Protein-enriched soup group (Experimental): Protein-enriched soup /day for use as a supplement with meals and strength training /week
  Interventions: Other: protein-enriched soup

INTERVENTIONS:
Other: protein-enriched soup — The participants in experimental group have a protein-enriched soup a day and do exercise a week
  Arms: Protein-enriched soup group

SUMMARY:
To evaluate the effects of protein-enriched soup plus exercise on muscle mass and muscle strength.

Besides, the investigators use the valued-based healthcare standard set as well as the Center for Epidemiological Studies-Depression, Charlson's comorbidity index Montreal Cognitive Assessment , and Mini Nutritional Assessment as outcome measures and to use the trial in validate additional supplement protein-enriched soup plus exercise could improve the vitality and health of mid-aged and old adults.

DETAILED DESCRIPTION:
With aging, functions of every organs become to decline. Muscle mass, is one of the decline. According to previous research, adults would lose 40% among from aged 20 to 70. If muscle mass decline combining with the decline of muscle strength is so called Sarcopenia.When muscle mass decline, infectious risk gets higher, and resilience after illness gets lower. In addition, activity and life quality are also responsible for falling, cognitive difficulty, disability and mortality among seniors. We hope to find out the etiologies of Sarcopenia through this program and develop prevention strategy and model to mollify the the negative effect of rapid aging society.

ELIGIBILITY:
Inclusion Criteria:

1. People who aged 50-75 years
2. Patients with following characteristics:
3. feeling loss in activity
4. detecting decline in self's walking speed.
5. feeling tired of doing everything.
6. having fell in last year.
7. People willing to follow the program and cooperate with us for following tracking.
8. People who are neither vegan nor vegetarian
9. People agree and be able to sign the informed consent.
10. the protein of the daily meal are less than 1.0g/kg

Exclusion Criteria:

1. People cannot intake provided meals (e.g.: vegans or vegetarians) or any other who is allergic to our diets.
2. People with any disease affecting their limbs, including:
3. having fracture on limbs in the past 6 months
4. having severe arthritis in the past 6 months
5. any other whom PI recognized as weak control of their nervous system( e.g.: Parkinson's disease and stroke).
6. People with intermittent limp caused by peripheral artery diseases
7. People with weak control of mental disorder
8. People with weak control of Cardiopulmonary disease
9. People with weak control of Malignant tumor
10. People with weak control of kidney diseases (eGFR <60ml/min/1.73)
11. People with Visual impairment and Hearing disorder which cannot help to complete the program.
12. People who have underwent hormone treatment and planned to undergo hormone treatment during program session.
13. Any other condition that PI recognized as not suitable

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline physical function after 12 weeks | baseline, 4, 12 weeks
  measured by hand grip, 6-minute walk distance, six-meter walking speed, 5 times sit-to-stand

SECONDARY OUTCOMES:
Change from baseline numbers of Complete blood count after 12 weeks | baseline, 4, 12 weeks
  Change from baseline numbers of Complete blood count after 12 weeks
Change from baseline concentration of Albumin after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of Albumin after 12 weeks
Change from baseline concentration of Alanine Aminotransferase (ALT) after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of Alanine Aminotransferase (ALT) after 12 weeks
Change from baseline concentration of Aspartate Aminotransferase (AST) after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of Aspartate Aminotransferase (AST) after 12 weeks
Change from baseline concentration of blood urea nitrogen after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of blood urea nitrogen after 12 weeks
Change from baseline concentration of Creatinin after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of Creatinin after 12 weeks
Change from baseline concentration of Fasting glucose after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of Fasting glucose after 12 weeks
Change from baseline concentration of Fasting insulin after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of Fasting insulin after 12 weeks
Change from baseline concentration of high-sensitivity C-reactive protein after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of high-sensitivity C-reactive protein after 12 weeks
Change from baseline concentration of 25-(OH)-Vit. D after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of 25-(OH)-Vit. D after 12 weeks
Change from baseline concentration of Leptin after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of Leptin after 12 weeks
Change from baseline concentration of urine protein after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of urine protein after 12 weeks
Changes form baseline QUALITY OF LIFE after 12 weeks | baseline, 4, 12 weeks
  measured by the 36-Item Short Form Health Survey (SF-36), ranged 0-100, higher values represent a better condition
Change from baseline Nutrition intake after 12 weeks | baseline, 4, 12 weeks
  measured by Mini-nutritional assessment questionnaire. ranged 0-30, higher values represent a better condition
Change from baseline depression after 12 weeks | baseline, 4, 12 weeks
  measured by the Center for Epidemiological Studies-Depression (CES-D) ranged 0-60, higher values represent a worse condition
Change from baseline cognitive ability after 12 weeks | baseline, 4, 12 weeks
  measured by Montreal Cognitive Assessment (MoCA) , ranged 0-30, higher values represent a better condition
Change from baseline body composition analysis after 12 weeks | baseline, 4, 12 weeks
  measured by RASM
Change from baseline concentration of Total Cholesterol after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of Total Cholesterol after 12 weeks
Change from baseline concentration of Triglyceride after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of Triglyceride after 12 weeks
Change from baseline concentration of high-density lipoprotein cholesterol after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of high-density lipoprotein cholesterol after 12 weeks
Change from baseline concentration of low-density lipoprotein cholesterol after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of low-density lipoprotein cholesterol after 12 weeks
Change from baseline concentration of dehydroepiandrosterone after 12 weeks | baseline, 4, 12 weeks
  Change from baseline concentration of dehydroepiandrosterone after 12 weeks
Change in International Physical Activity Questionnaire (IPAQ) after 12 weeks | baseline, 4, 12 weeks
  Change in physical activity measured by IPAQ, indicates that spent being physically active thin the prior 7 days.There are no established thresholds for presenting MET-minutes, the IPAQ Research Committee proposes that reported as comparisons of median values and interquartile ranges for different populations from baseline to 12 weeks in all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, MD.PhD., Principal Investigator — Center for Healthy Longevity and Aging Sciences, National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan